CLINICAL TRIAL: NCT03707392
Title: Quality Outcomes of Ostomy Teaching: A Randomized Trial of Inpatient Stoma-Nurse Teaching Versus Stoma Teaching Video Combined With Inpatient Stoma-Nurse Teaching
Brief Title: A Randomized Trial of Inpatient Stoma-Nurse Teaching Versus Stoma Teaching Video Combined With Inpatient Stoma-Nurse Teaching
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sang Won Lee, Professor of Clinical Surgery, Chief, Division of Colorectal Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-17-00982
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Ileostomy - Stoma; Colostomy Stoma
Keywords: stoma education

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard preoperative and postoperative stoma teaching including ostomy nurse teaching and educational materials
  Interventions: Other: Control - Standard ostomy education
- Treatment (Experimental): Ostomy care educational video combined with standard preoperative and postoperative stoma teaching including ostomy nurse teaching and educational materials
  Interventions: Other: Ostomy Education Video

INTERVENTIONS:
Other: Ostomy Education Video — Ostomy education video in addition to standard ostomy education including preoperative and postoperative ostomy nurse teaching and educational materials
  Arms: Treatment
Other: Control - Standard ostomy education — Standard ostomy education including preoperative and postoperative ostomy nurse teaching and educational materials
  Arms: Control

SUMMARY:
Adult patients without prior history of ostomy, undergoing elective surgery involving a new ileostomy or colostomy will be randomized to receive standard ostomy nurse teaching or ostomy nurse teaching combined with preoperative and postoperative stoma care teaching video. Post operative outcomes including delay in discharge and stoma-related complications will be tracked.

DETAILED DESCRIPTION:
Adult patients without prior history of ostomy, undergoing surgery involving a new ileostomy or colostomy will be randomized to receive standard ostomy nurse teaching or ostomy nurse teaching combined with preoperative and postoperative stoma care teaching video. Patients will be consented and randomized at the time of preoperative clinic visit. All patients will receive standard preoperative ostomy teaching materials and education from the surgeon and clinic nurse. Patients randomized to the treatment arm will receive additional take-home teaching materials based on the American College of Surgeons Ostomy Teaching videos.

After post-operative inpatient ostomy-nurse teaching, and prior to discharge from the hospital, patients will fill out a survey detailing their level of comfort with various aspects of ostomy home care. Patients in the treatment arm will be be asked to review the ostomy teaching videos and fill out the survey prior to discharge. Primary outcome will be delay in discharge from hospital due to stoma-teaching related issues. Secondary outcomes will include rate of calls to the clinic for stoma-related questions, stoma-related clinic/urgent care/emergency department visits, and stoma-related complications.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 yrs of age
* undergoing elective surgery including plan for ileostomy or colostomy

Exclusion Criteria:

* patients unable or unwilling to provide informed consent for any reason, including patients with inadequate capacity for decision making.
* Patients undergoing emergent surgery
* Vulnerable populations such as prison and psychiatric ward patients
* Patients who for any reason do not undergo construction of pre-operatively planned stoma
* Patients with history of previous stoma creation
* Patients who are not their own primary caregivers will also be excluded, including those patients who are planned to be discharged to care facility or nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Delay in hospital discharge | through initial inpatient hospital stay: an average of 5 days
  Delay in hospital discharge due to need for additional ostomy teaching

SECONDARY OUTCOMES:
Length of stay | through initial inpatient hospital stay: an average of 5 days
  overall length of inpatient hospitalization
Hospital Readmission | within 30 days, and within 30-60 days postoperatively
  rate of readmission to hospital after surgery
Phone Calls | within 60 days of discharge
  Number of phone calls to surgical team after discharge
Clinic/Urgent Care/Emergency Department visits | within 60 days of discharge
  number of Clinic/Urgent Care/Emergency Department visits

CONTACTS AND LOCATIONS:
Overall Officials: Sang W Lee, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD